

## **PARTICIPANT CONSENT FORM**

## The SToICAL Study – The Soft Tissue Injection of Corticosteroid And Local anaesthetic

| Name of Researcher: Mr C Goz | zard/ Miss S Fullilove/ Dr E Doyl | rle/ Mr M Jones/ Mr J Evans |
|---|---|---|
| Patient participation number: | | |
| Study treatment number: | | |
| | | Please initial all boxes |
| 1. I confirm that I have read a | nd understand the patient informa | ation sheet dated |
| , | (version) for the above study. I have had the opportunity to consider the | |
| information, ask questions and have had these answered satisfactorily. | | |
| 2. I understand that my partic | ipation is voluntary and that I am | n free to withdraw at any time |
| without giving any reason, without my medical care or legal rights being affected. | | |
| | | _ |
| | , | |
| may be looked at by individuals from regulatory authorities or from the NHS Trust, where it is | | |
| relevant to my taking part in this research. I give permission for these individuals to have access to my records. | | |
| addeds to my records. | | _ |
| 4. I agree to be contacted by a member of the study team as part of the study follow-up the day | | |
| after my steroid injection | | |
| 5. I agree to my GP being info | rmed of my participation in the si | tudy |
| 5. Tagree to my Gr being into | imed of my participation in the si | luuy. |
| 6. I agree to take part in the above study. | | |
| | | L |
| 7. I would like to be informed of the results of the study, when they are available and agree that my contact details can be retained for this purpose. | | |
| contact details can be retail | ined for tine purpose. | L |
| Name of Participant | Date | Signature |
| Name of Person taking consent | Date | Signature |
| When completed: 1 copy for part original copy for researcher site | | 1 copy provided to the sponsor and |

IRAS No:259336